CLINICAL TRIAL: NCT04626375
Title: Effects of L-arginine on Myocardial Energetic Efficiency and Global Longitudinal Strain
Acronym: BIOCARDIO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: Prof. Raffaele Izzo (Unknown); Prof. Costantino Mancusi (Unknown)
Responsible Party: Principal Investigator, Bruno Trimarco, Full Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BIOARGININA
Record Dates: First submitted 2020-02-16; First posted 2020-11-12 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Myocardial Dysfunction
Keywords: Hypertension; Echocardiography; Global Longitudinal Strain
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (2 vials per os without active substance every 12 hours)
  Interventions: Drug: Placebo oral tablet
- Bioarginine (Active Comparator): Bioarginine (2 vials per os of 1.66 g every 12 hours)
  Interventions: Drug: Bioarginine

INTERVENTIONS:
Drug: Bioarginine — In the Bioarginine group the partecipants take bioarginine (2 vials per os of 1.66 g every 12 hours) for 4 week
  Arms: Bioarginine
Drug: Placebo oral tablet — In the Placebo group the participants take bio-arginine (2 vials per os of 1.66 g every 12 hours) for 4 week
  Arms: Placebo

SUMMARY:
The study is designed to evaluate the effects of L-arginine on myocardial structure and function and circulating microRNAs in patients with arterial hypertension.

The study will analyze the impact of 4 weeks treatment randomized to L-arginine or placebo, on mechanical-energy efficiency (MEE) and longitudinal strain in patients with arterial hypertension. The investigators will also assess whether the changes in MEE and strain induced by L-arginine treatment is associated with changes in circulating micro RNAs.

DETAILED DESCRIPTION:
The patients and controls will be recruited at the Hypertension research center of Federico II university hospital.

The overall duration of the study will be 4 weeks for each participant. Blood pressure, heart rate, echocardiogram and blood sample will be collected for each patients at randomization and after 4 weeks of treatment.

Patients or controls will be randomized to receive bioarginine (up to 2 vials per os of 1.66 g every 12 hours) or placebo (up to 2 vials per os without active substance every 12 hours). Before the start of treatment, patients will receive a peripheral venous blood sample (10-12 ml), which will be identified through the use of an alphanumeric code (PRE-XXXYYY). In addition, patients will undergo full echocardiographic examination (the parameters will be reported in a password-protected database, using the same identification codes used for blood sampling). The duration of the treatment will be 4 weeks. At the end of the treatment, the patients will receive a peripheral venous blood sample (10-12 ml) which will be identified through the use of an alphanumeric code (POST-XXXYYY) and full echocardiographic examination.

In some controls, we will run an explorative study to verify the eventual impact of Bioarginine on standardized physical exercise. Healthy controls will undergo a physical exercise according to their preference, at baseline and after 4 weeks of treatment or placebo. Ear lobe blood samples are taken before and after the effort and analyzed for serum lactate content using the reflectance photometric enzymatic reaction method. All L-arginine and placebo, made up of the L-arginine vehicle without the active substance, will be offered free of charge by the Farmaceutici DAMOR company.

ELIGIBILITY:
Inclusion Criteria:

* Low values of mechanical-energy efficiency
* Sinus rhytm

Exclusion Criteria:

* Atrial fibrillation
* Taking Beta blockers
* Pregnancy
* Cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Myocardial Energetic Efficiency | 4 week
  Myocardial Energetic Efficiency is calculated as SV/HR/60/LV mass measuring the amount of blood pumped by left ventricle each second per each gram of left ventricular mass
Change in global longitudinal strain | 4 week
  Global longitudinal strain represent the longitudinal shortening as a percentage (change in length as a proportion to baseline length) (%)

SECONDARY OUTCOMES:
Variation of circulating non-coding RNA | 4 week
  Variation of circulating non-coding RNA is evaluated by blood samples of venous blood and expressed as fold change to placebo patients

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Trimarco, MF, Study Director — Federico II University, DPT of Advanced Biomedical Sciences
Locations (1):
- Ambulatorio Ipertensione e Unità Coronarica Federico II University, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shah AM, Solomon SD. Myocardial deformation imaging: current status and future directions. Circulation. 2012 Jan 17;125(2):e244-8. doi: 10.1161/CIRCULATIONAHA.111.086348. No abstract available. PMID 22249531
- [Result] Karlsen S, Dahlslett T, Grenne B, Sjoli B, Smiseth O, Edvardsen T, Brunvand H. Global longitudinal strain is a more reproducible measure of left ventricular function than ejection fraction regardless of echocardiographic training. Cardiovasc Ultrasound. 2019 Sep 2;17(1):18. doi: 10.1186/s12947-019-0168-9. PMID 31477137
- [Result] Tschope C, Senni M. Usefulness and clinical relevance of left ventricular global longitudinal systolic strain in patients with heart failure with preserved ejection fraction. Heart Fail Rev. 2020 Jan;25(1):67-73. doi: 10.1007/s10741-019-09853-7. PMID 31489515
- [Result] Bianco CM, Farjo PD, Ghaffar YA, Sengupta PP. Myocardial Mechanics in Patients With Normal LVEF and Diastolic Dysfunction. JACC Cardiovasc Imaging. 2020 Jan;13(1 Pt 2):258-271. doi: 10.1016/j.jcmg.2018.12.035. Epub 2019 Jun 12. PMID 31202770
- [Result] Nahum J, Bensaid A, Dussault C, Macron L, Clemence D, Bouhemad B, Monin JL, Rande JL, Gueret P, Lim P. Impact of longitudinal myocardial deformation on the prognosis of chronic heart failure patients. Circ Cardiovasc Imaging. 2010 May;3(3):249-56. doi: 10.1161/CIRCIMAGING.109.910893. Epub 2010 Mar 16. PMID 20233858
- [Result] Kalam K, Otahal P, Marwick TH. Prognostic implications of global LV dysfunction: a systematic review and meta-analysis of global longitudinal strain and ejection fraction. Heart. 2014 Nov;100(21):1673-80. doi: 10.1136/heartjnl-2014-305538. Epub 2014 May 23. PMID 24860005